CLINICAL TRIAL: NCT01503164
Title: Sleep, Obesity, and Metabolism in Normal and Overweight Subjects: Effects of CPAP on Glucose Metabolism
Brief Title: Effects of Continuous Positive Airway Pressure (CPAP) on Glucose Metabolism
Acronym: SOMNOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00036672; 2R01HL075078 (NIH)
Record Dates: First submitted 2011-12-29; First posted 2012-01-02 (Estimated); Results first posted 2017-10-19 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Obstructive Sleep Apnea; Sleep Apnea; Sleep-disordered Breathing
Keywords: Obstructive sleep apnea; Sleep Apnea; Sleep-disordered breathing; Insulin sensitivity; Glucose tolerance; Type 2 diabetes
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Insulin Resistance; Diabetes Mellitus, Type 2 | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Positive pressure therapy (PAP) (Active Comparator): Positive airway pressure(PAP) therapy is the standard of care for patients with obstructive sleep apnea. During sleep, a mask is worn over the nose and connected to the PAP machine.
  Interventions: Device: Positive Pressure Therapy (PAP)
- Lifestyle counseling (Sham Comparator)
  Interventions: Behavioral: LifeStyle Counseling

INTERVENTIONS:
Device: Positive Pressure Therapy (PAP) — Positive pressure therapy is the standard of care for managing obstructive sleep apnea. It entails wearing a mask that is connected to the PAP device which deliver pressure to the upper airway during sleep.
  Other Names: CPAP
  Arms: Positive pressure therapy (PAP)
Behavioral: LifeStyle Counseling — Subjects randomized to the lifestyle (and nutritional) counseling arm will be given advice on a balanced dietary and exercise plan.
  Other Names: Dietary and Lifestyle Counseling
  Arms: Lifestyle counseling

SUMMARY:
Obstructive sleep apnea affects approximately 2-4% of middle-aged adults in the general population and is associated with several medical conditions including hypertension and coronary artery. Research over the last decade has shown that obstructive sleep apnea may also increase the propensity for insulin resistance, glucose intolerance, and type 2 diabetes mellitus. Positive airway pressure (PAP) is the first line therapy for the treatment of obstructive sleep apnea. While PAP therapy has several favorable effects such as improvements in daytime sleepiness and quality of life, it is not clear whether using PAP therapy can alter metabolic risk. The overall objective of this study is to examine whether treatment of obstructive sleep apnea with positive airway pressure therapy improves glucose tolerance and insulin sensitivity. The primary hypothesis of this study is that PAP therapy of obstructive sleep apnea will improve in insulin sensitivity and glucose metabolism.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus is one of the most prevalent medical conditions, affecting a staggering 246 million people worldwide. Obstructive sleep apnea is a relatively common and often undiagnosed condition in the general population. Cross-sectional studies of clinic and population-based samples suggest that up to 40% of patients with obstructive sleep apnea have type 2 diabetes and up to 75% of patients with type 2 diabetes have obstructive sleep apnea. There is increasing evidence that the pathophysiological features of intermittent hypoxia and sleep fragmentation may be responsible for altering glucose homeostasis and worsening insulin sensitivity. The mechanisms through which obstructive sleep apnea impairs glucose metabolism are largely unknown. While intermittent hypoxemia and sleep fragmentation are likely to play an essential role, the relative contribution of each in the causal pathway remains to be determined. Moreover, whether the adverse effects of intermittent hypoxia and sleep fragmentation are mediated through an increase in sympathetic nervous system activity, alterations in corticotropic function, and/or systemic inflammation is not known. Furthermore, it remains to be determined whether positive pressure therapy for obstructive sleep apnea has salutary effects on glucose metabolism. Many of the available studies examining the effects of PAP on glucose tolerance and insulin sensitivity are plagued by small sample sizes, lack of a control group, and limited data on compliance with positive pressure therapy. The current study will assess, using a community-based sample, whether treatment of obstructive sleep apnea with positive pressure therapy will improve insulin sensitivity, as assessed by the frequently sample intravenous glucose tolerance test (primary outcome measure).

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Obstructive sleep apnea (untreated)
* Ability to comply with study-related assessments

Exclusion Criteria:

* Inability to consent or commit to the required visits
* Diabetes mellitus (fasting glucose > 126 mg/dl)
* Use of insulin or oral hypoglycemic agent
* Weight change of 10% in last six months
* Use of oral steroids in the last six months
* Severe pulmonary disease (i.e., COPD)
* Renal or hepatic insufficiency
* Recent Myocardial Infarction (MI) or stroke (< 3 months)
* Occupation as a commercial driver
* Active substance use
* Untreated thyroid disease
* Pregnancy
* Anemia (Hematocrit < 30%)
* Any history of seizures or other neurologic disease
* Poor sleep hygiene or sleep disorder other than sleep apnea
* Excessive subjective sleepiness (Epworth score > 18)

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naresh M Punjabi, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Young T, Peppard PE, Gottlieb DJ. Epidemiology of obstructive sleep apnea: a population health perspective. Am J Respir Crit Care Med. 2002 May 1;165(9):1217-39. doi: 10.1164/rccm.2109080. PMID 11991871
- [Background] Punjabi NM, Ahmed MM, Polotsky VY, Beamer BA, O'Donnell CP. Sleep-disordered breathing, glucose intolerance, and insulin resistance. Respir Physiol Neurobiol. 2003 Jul 16;136(2-3):167-78. doi: 10.1016/s1569-9048(03)00079-x. PMID 12853008
- [Background] Tasali E, Mokhlesi B, Van Cauter E. Obstructive sleep apnea and type 2 diabetes: interacting epidemics. Chest. 2008 Feb;133(2):496-506. doi: 10.1378/chest.07-0828. PMID 18252916
- [Background] Punjabi NM; Workshop Participants. Do sleep disorders and associated treatments impact glucose metabolism? Drugs. 2009;69 Suppl 2:13-27. doi: 10.2165/11531150-000000000-00000. PMID 20047348
- [Derived] Aurora RN, Swartz R, Punjabi NM. Misclassification of OSA severity with automated scoring of home sleep recordings. Chest. 2015 Mar;147(3):719-727. doi: 10.1378/chest.14-0929. PMID 25411804

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Positive Pressure Therapy (PAP) | Lifestyle Counseling
Started | 55 | 56
Completed | 53 | 55
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: 55 randomized to PAP (2 dropout); 56 randomized to lifestyle (1 dropout)
Groups:
- Lifestyle Counseling: Positive Pressure Therapy (PAP): Positive pressure therapy is the standard of care for managing obstructive sleep apnea. It entails wearing a mask that is connected to the PAP device which deliver pressure to the upper airway during sleep.
  LifeStyle Counseling: Subjects randomized to the lifestyle (and nutritional) counseling arm will be given advice on a balanced dietary and exercise plan.
- Total: Total of all reporting groups
Arm/Group | Positive Pressure Therapy (PAP) | Lifestyle Counseling | Total
Number analyzed (Participants) | 53 | 55 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 44 | 89
  >=65 years | 8 | 11 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (9.2) | 57.2 (8.2) | 56.0 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 41 | 39 | 80
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53 | 55 | 108

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity (SI)
Description: Insulin sensitivity will be determined with the insulin-modified frequently sampled intravenous glucose tolerance test (IVGTT) before and 2-months after study intervention. This test requires administration of a weight-adjusted dose of D50W as an IV bolus at time "zero". After the glucose bolus, blood samples are drawn at the scheduled times for 3-hours. At the 20-minute mark, a weight-adjusted dose of regular insulin is administered. The resulting serum is analyzed for glucose and insulin and the "minimal model" (MINMOD) will be used to derive insulin sensitivity. A low SI signifies low insulin sensitivity and high SI represents high insulin sensitivity.
Time Frame: Baseline
Population: 55 randomized to PAP (2 dropout); 56 randomized to lifestyle (1 dropout)
Measure: Mean (Standard Deviation); unit: [mU/L]^-1 x [min]^-1
Arm/Group | Positive Pressure Therapy (PAP) | Lifestyle Counseling
Number analyzed (Participants) | 53 | 55
[mU/L]^-1 x [min]^-1 | 1.95 (1.21) | 2.22 (1.45)

2. Primary Outcome: Insulin Sensitivity (SI)
Description: as for outcome 1
Time Frame: 2 months after intervention
Population: 55 randomized to PAP (2 dropout); 56 randomized to lifestyle (1 dropout)
Measure: Mean (Standard Deviation); unit: [mU/L]^-1 x [min]^-1
Arm/Group | Positive Pressure Therapy (PAP) | Lifestyle Counseling
Number analyzed (Participants) | 53 | 55
[mU/L]^-1 x [min]^-1 | 3.01 (2.77) | 1.83 (1.03)

3. Secondary Outcome: Glucose Effectiveness (SG)
Description: Glucose effectiveness is the ability for glucose to move intracellularly in the absence of insulin. It is a parameter that results from the MINMOD analysis of the serum glucose and insulin levels derived from the frequently sampled intravenous glucose tolerance test. Low SG indicates a lower predisposition for glucose disposal independent of any effects of insulin.
Time Frame: Baseline
Population: 55 randomized to PAP (2 dropout); 56 randomized to lifestyle (1 dropout)
Measure: Mean (Standard Deviation); unit: [min]^-1
Arm/Group | Positive Pressure Therapy (PAP) | Lifestyle Counseling
Number analyzed (Participants) | 53 | 55
[min]^-1 | 0.01498 (0.006408) | 0.01537 (0.00636)

4. Secondary Outcome: Glucose Effectiveness (SG)
Description: as for outcome 3
Time Frame: 2 months after intervention
Population: 55 randomized to PAP (2 dropout); 56 randomized to lifestyle (1 dropout)
Measure: Mean (Standard Deviation); unit: [min]^-1
Arm/Group | Positive Pressure Therapy (PAP) | Lifestyle Counseling
Number analyzed (Participants) | 53 | 55
[min]^-1 | 0.01720 (0.01094) | 0.01385 (0.00636)

5. Secondary Outcome: Disposition Index (DI)
Description: The disposition index is the mathematical product of insulin sensitivity (SI) and acute insulin response to glucose (AIRG) both of which are derived from the MINMOD analysis of the frequently sampled intravenous glucose tolerance test data. A low DI is indicative of a higher risk of developing diabetes.
Time Frame: Baseline
Population: 55 randomized to PAP (2 dropout); 56 randomized to lifestyle (1 dropout)
Measure: Mean (Standard Deviation); unit: [mU/L]^-1 x [min]^-1] x [mU/L-min]
Arm/Group | Positive Pressure Therapy (PAP) | Lifestyle Counseling
Number analyzed (Participants) | 53 | 55
[mU/L]^-1 x [min]^-1] x [mU/L-min] | 931.4 (957.1) | 1093.1 (1037.9)

6. Secondary Outcome: Disposition Index (DI)
Description: The disposition index is the mathematical product of insulin sensitivity (SI) and acute insulin response to glucose (AIRG) both of which are derived from the MINMOD analysis of the frequently sampled intravenous glucose tolerance test data.
Time Frame: 2 months after intervention
Population: 55 randomized to PAP (2 dropout); 56 randomized to lifestyle (1 dropout)
Measure: Mean (Standard Deviation); unit: [mU/L]^-1 x [min]^-1] x [mU/L-min]
Arm/Group | Positive Pressure Therapy (PAP) | Lifestyle Counseling
Number analyzed (Participants) | 53 | 55
[mU/L]^-1 x [min]^-1] x [mU/L-min] | 1385.9 (1670.1) | 815.4 (579.5)

7. Secondary Outcome: Acute Insulin Response to Glucose (AIRG)
Description: The acute insulin response to glucose (AIRG) value is derived from the MINMOD analysis of the glucose and insulin levels obtained during the frequently sampled intravenous glucose tolerance test. A low AIRG indicates decreased ability of the pancreas to secrete insulin.
Time Frame: Baseline
Population: 55 randomized to PAP (2 dropout); 56 randomized to lifestyle (1 dropout)
Measure: Mean (Standard Deviation); unit: [mU/L-min]
Arm/Group | Positive Pressure Therapy (PAP) | Lifestyle Counseling
Number analyzed (Participants) | 53 | 55
[mU/L-min] | 537.48 (394.88) | 632.38 (728.65)

8. Secondary Outcome: Acute Insulin Response to Glucose (AIRG)
Description: as for outcome 7
Time Frame: 2 months after intervention
Population: 55 randomized to PAP (2 dropout); 56 randomized to lifestyle (1 dropout)
Measure: Mean (Standard Deviation); unit: [mU/L-min]
Arm/Group | Positive Pressure Therapy (PAP) | Lifestyle Counseling
Number analyzed (Participants) | 53 | 55
[mU/L-min] | 513.06 (338.41) | 563.64 (546.20)

9. Secondary Outcome: Endothelial Function
Description: Endothelial function will be assessed using peripheral arterial tonometry using the Endo-PAT device. Using the EndoPat device, the relative vasoconstriction of occluded versus non-occluded arms was derived and provided the relative hyperemic index.
Time Frame: Baseline
Population: Data was unable to be collected for all participants in this outcome measure.
Measure: Mean (Standard Deviation); unit: ratio of occluded versus non-occluded
Arm/Group | Positive Pressure Therapy (PAP) | Lifestyle Counseling
Number analyzed (Participants) | 49 | 54
ratio of occluded versus non-occluded | 1.91 (0.46) | 1.92 (0.49)

10. Secondary Outcome: Endothelial Function
Description: as for outcome 9
Time Frame: 2 month after intervention
Population: Data was not collected for all participants for this outcome measure. Participants for whom data was available are included in analysis.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Positive Pressure Therapy (PAP) | Lifestyle Counseling
Number analyzed (Participants) | 49 | 54
ratio | 1.90 (0.53) | 1.91 (0.46)

11. Secondary Outcome: Area Under the Curve Assessed by Oral Glucose Tolerance Test
Description: Results of the oral glucose tolerance test will be analyzed using indices derived from the serial glucose and insulin levels over the 2 hour period. This will be the area under the glucose/ insulin curves
Time Frame: Baseline
Population: 55 randomized to PAP (2 dropout); 56 randomized to lifestyle (1 dropout)
Measure: Mean (Standard Deviation); unit: mg/dL per 120 min
Arm/Group | Positive Pressure Therapy (PAP) | Lifestyle Counseling
Number analyzed (Participants) | 53 | 55
mg/dL per 120 min | 7939.9 (3327.8) | 7245.31 (2988.4)

12. Secondary Outcome: Area Under the Curve Assessed by Oral Glucose Tolerance Test (OGTT)
Description: Results of the oral glucose tolerance test will be analyzed using indices derived from the serial glucose and insulin levels over a 2 hour period 2 months post intervention. This will be the area under the glucose/ insulin curves
Time Frame: 2 month after intervention
Population: 55 randomized to PAP (2 dropout); 56 randomized to lifestyle (1 dropout)
Measure: Mean (Standard Deviation); unit: mg/dL per 120 min
Arm/Group | Positive Pressure Therapy (PAP) | Lifestyle Counseling
Number analyzed (Participants) | 53 | 55
mg/dL per 120 min | 7531.8 (3179.2) | 7655.1 (3057.6)

ADVERSE EVENTS:
Time Frame: up to 4 months after enrollment in study
Arm/Group | Positive Pressure Therapy (PAP) | Lifestyle Counseling
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/56
Other Adverse Events (participants affected / at risk) | 0/55 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes